CLINICAL TRIAL: NCT04812405
Title: Assessment of the Difference of Fluoresce of the TRIOS 4 Intraoral Scanner of the Same Surface at In Vivo and In Vitro Conditions
Brief Title: Automated Caries Detection Using a 3D Intraoral Scanner. An in Vivo Validation Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Rahiotis Chris, Associate Professor, National and Kapodistrian University of Athens
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 385
Record Dates: First submitted 2021-03-18; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Healthy Patients
Keywords: caries detection; in vivo; intraoral scanner; ICDAS; histology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Teeth (Other): Occlusal examination
  Interventions: Diagnostic Test: Trios4

INTERVENTIONS:
Diagnostic Test: Trios4 — Examination of occlusal surfaces with 3D scanner and optical criteria
  Other Names: ICDAS

SUMMARY:
This in vivo study with in vitro validation assessed four different algorithms (ALG1-ALG4) implemented in the intraoral scanner system for automated caries detection and classification. 3D scans of the examined teeth were obtained both in vivo and vitro, i.e. before and after tooth extraction, in order to assess any possible differences in the performance of the algorithms at different conditions. The latter could potentially help drawing some conclusions regarding i) the validity of the in vitro studies assessing fluorescence method for caries detection, and ii) the in vivo applicability of in vitro results obtained in the past and the future. Additionally, visual-tactile examination using the ICDAS (ICDAS II) criteria19 was conducted on the same teeth in vivo and histological assessment was used as reference test in vitro.

ELIGIBILITY:
Inclusion Criteria:

* Patients with permanent molars / premolars,
* Sound teeth or with caries lesions on the occlusal surfaces.

Exclusion Criteria:

* Front teeth / deciduous teeth
* Teeth with fillings
* Teeth with broken crown
* Teeth with extensive lesions on the lateral surfaces.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2020-06-03 (Actual); Primary Completion 2020-11-15 (Actual); Study Completion 2021-03-10 (Actual)

PRIMARY OUTCOMES:
Agreement of In vivo validation with in vitro caries detection | 1 year
  To assess the difference in vivo and in vitro the fluorescence emitted of the TRIOS FLUO intraoral scanner from occlusal surface from 3rd molar before and after extraction

CONTACTS AND LOCATIONS:
Locations (1):
- Dentistry, Athens, Greece

IPD SHARING:
Plan to Share IPD: No